CLINICAL TRIAL: NCT03990389
Title: Automated Symptom Tracking for Measurement-Based Care of Depression
Brief Title: Tracking Depression Symptoms With a Health Chatbot
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Chicago (Other)
Collaborators: Endeavor Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB16-1802
Record Dates: First submitted 2019-03-13; First posted 2019-06-19 (Actual); Results first posted 2022-05-12 (Actual); Last update posted 2022-05-12 (Actual); Status verified 2022-04

CONDITIONS: Depression, Postpartum; Depression, Unipolar
MeSH Terms: conditions — Depression, Postpartum; Depressive Disorder

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (3):
- Usual Care Group (No Intervention): Subjects will undergo screening including Rapid Estimate of Adult Literacy in Medicine (REALM-R) and Edinburgh Postnatal Depression Scale (EPDS) and a few additional questions.
  Eligible subjects randomized to usual care will receive monthly reminder phone calls from a research coordinator. Subjects will receive an email with a link to surveys for the purpose of collecting information on depression severity, medication adherence, self-efficacy, side-effect burden, and maternal functioning.
  All participants will be asked to participate in a semi-structured debrief interview upon study completion.
- Chabot Care Group (Experimental): Subjects will undergo screening including REALM-R and EPDS and a few additional questions.
  Eligible subjects randomized to chatbot care will receive monthly reminder phone calls from a research coordinator. Subjects will receive an email with a link to surveys for the purpose of collecting information on depression severity, medication adherence, self-efficacy, side-effect burden, and maternal functioning.
  In addition to the above procedures, eligible subjects randomized to chatbot care will receive weekly messages from the chatbot asking them to complete a depression severity measure and side-effect burden assessments. Within week 1 subjects will receive a check-in call from a study coordinator to answer any questions regarding use of the chatbot.
  All participants will be asked to participate in a semi-structured debrief interview upon study completion.
  Interventions: Device: Chatbot Intervention
- Provider Subject Cohort (No Intervention): 20 provider subjects from each study site will be enrolled to ensure they understand the study and consent to have their patients enrolled in the study

INTERVENTIONS:
Device: Chatbot Intervention — a chatbot will be used to monitor depression severity
  Arms: Chabot Care Group

SUMMARY:
The goal of this research is to bridge a significant "effectiveness" gap in the treatment of depression. The investigators have developed a chatbot which will assist in performing measurement-based care (MBC) via Facebook Messenger. Participants will be randomized to either Usual Care or Usual Care with additional Chatbot Care.

DETAILED DESCRIPTION:
The goal of this research is to bridge a significant "effectiveness" gap in the treatment of depression. The investigators will be looking specifically at depressed women soon after they give birth, otherwise known as known as perinatal depression. Measurement-based care (MBC) which involves the use of quantitative assessments for depression screening, diagnosis, and symptom monitoring is recognized as one of the keys to depression management. MBC can be difficult to implement within the clinical setting due to the administrative overhead and close follow-up required. It is reasonable to hypothesize that low rates of MBC adoption are responsible for low rates of adequate depression care.

The investigators have developed an automated conversational agent or "chatbot" (CB) for delivering MBC via Facebook Messenger. The investigators hypothesize that the use of CB-MBC, which combines a conversational interface with state-of-the-art quantitative assessments, will improve depression symptom severity for patients with perinatal depression. If successful, this project will provide primary care physicians with a new and inexpensive method for delivering better and safer care to their patients with depression. This study works to determine the impact of the chatbot in improving depression outcomes for patients under treatment for perinatal depression.

ELIGIBILITY:
Inclusion Criteria:

* Provider Subject Cohort: residents and attendings from University of Chicago Medical Center OBGYN and NorthShore Hospital OBGYN clinics.
* Patient Subject Cohort:

  1. Age ≥ 18 years and able to and demonstrate English reading literacy of at least 8th-grade level (REALM-R ≥ 6)
  2. Postnatal women newly diagnosed or receiving treatment for non-psychotic unipolar depression with a severity-based entry criterion of moderate to severe (EPDS ≥ 12)
  3. Willing to participate and able to give written informed consent
  4. Must own a smart phone with a data plan
  5. Must have a Facebook account and Facebook Messaging app on phone (or willing to create account/download app today)
  6. Sufficient cognitive ability to provide self-report data on a computer touchscreen/ standard computer with minimal assistance

Exclusion Criteria:

* Provider Subject Cohort: None
* Patient Subject Cohort:

  1. Subjects with documented dysthymia or Axis II diagnoses
  2. Subjects with self-reported or documented history of: anorexia or bulimia, obsessive compulsive disorder or prior hospitalization for suicidal ideation
  3. Active suicidality as determined by clinician
  4. Non-English speakers

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2019-02-20 (Actual); Primary Completion 2020-02-29 (Actual); Study Completion 2020-02-29 (Actual)

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - University of Chicago, Chicago, Illinois
  - NorthShore University HealthSystem, Skokie, Illinois

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Excluded Patient Subjects (n = 35)
  * EPDS < 12 (n = 12)
  * Spanish speaking only (n = 2)
  * No Facebook account (n=1)
  * Consent not returned (n=18)
  * Refused (n = 2)
  No data was collected for the providers as no results related to the providers were reported.
Groups:
- No Intervention: Usual Care Group: Subjects will undergo screening including Rapid Estimate of Adult Literacy in Medicine (REALM-R) and Edinburgh Postnatal Depression Scale (EPDS) and a few additional questions.
- Experimental: Chabot Care Group: Subjects will undergo screening including REALM-R and EPDS and a few additional questions.
Period: Overall Study
Arm/Group | No Intervention: Usual Care Group | Experimental: Chabot Care Group
Started | 15 | 16
Completed | 12 | 16
Not Completed | 3 | 0
Not completed — Lost to Follow-up | 3 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | No Intervention: Usual Care Group | Experimental: Chabot Care Group | Total
Number analyzed (Participants) | 15 | 16 | 31
Age, Continuous [Mean (Standard Deviation); unit: years] | 31.3 (4.4) | 33.1 (2.7) | 32.2 (3.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 16 | 31
  Male | 0 | 0 | 0
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Longitudinal Change in Depression Severity
Description: Measured by the Edinburgh Postnatal Depression Scale (EPDS) Range 0-30 (dimensionless) Risk of depression goes up with an increasing score
Time Frame: 3 months
Population: missing values at month 1, month 2, and month 3
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | No Intervention: Usual Care Group | Experimental: Chabot Care Group
Number analyzed (Participants) | 15 | 16
score on a scale
  baseline | 16.13 (1.17) | 14.06 (1.13)
  month 1: number analyzed (Participants) | 12 | 16
  month 1 | 10.47 (1.29) | 10.69 (1.13)
  month 2: number analyzed (Participants) | 11 | 14
  month 2 | 8.23 (1.33) | 11.35 (1.19)
  month 3: number analyzed (Participants) | 11 | 15
  month 3 | 9.64 (1.33) | 10.87 (1.16)
Statistical Analysis 1: Comparison: No Intervention: Usual Care Group vs Experimental: Chabot Care Group; Test type: Superiority; p = 0.0618, Mixed Models Analysis — Three degrees of freedom for the interaction test
Statistical Analysis 2: Comparison: No Intervention: Usual Care Group vs Experimental: Chabot Care Group; Test type: Superiority; p = 0.63, Mixed Models Analysis — Bonferroni correction for 3 times points; estimated treatment effect at month 1 = -2.29, Standard Error of Mean 1.8
Statistical Analysis 3: Comparison: No Intervention: Usual Care Group vs Experimental: Chabot Care Group; Test type: Superiority; p = 0.018, Mixed Models Analysis — Bonferroni correction for 3 times points; estimated treatment effect at month 2 = -5.19, Standard Error of Mean 1.9
Statistical Analysis 4: Comparison: No Intervention: Usual Care Group vs Experimental: Chabot Care Group; Test type: Superiority; p = 0.234, Mixed Models Analysis — Bonferroni correction for 3 times points; estimated treatment effect at month 3 = -3.30, Standard Error of Mean 1.9

2. Secondary Outcome: Change in Depression Severity
Description: Measured by the Computerized Adaptive Test-Depression Inventory (CAT-DI) and calculated change in Edinburgh Postnatal Depression Scale (EPDS) between Baseline and 3 months.
  Edinburgh Postnatal Depression Scale (EPDS) Range 0-30 (dimensionless) Risk of depression goes up with an increasing score
Time Frame: 3 months
Population: Four missing values in the Usual Care Group and one missing value in the Chabot Care Group
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | No Intervention: Usual Care Group | Experimental: Chabot Care Group
Number analyzed (Participants) | 11 | 15
score on a scale | -6.2 (4.3) | -3.1 (5.4)
Statistical Analysis 1: Comparison: No Intervention: Usual Care Group vs Experimental: Chabot Care Group; Test type: Other; p = 0.116, t-test, 2 sided

3. Secondary Outcome: Change in Side-effect Burden
Description: Measured by the Frequency, Intensity, and Burden of Side Effects Rating (FIBSER) questionnaire
Time Frame: 3 months
Population: No data collected
Arm/Group | No Intervention: Usual Care Group | Experimental: Chabot Care Group
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Change in Maternal Function
Description: Measured by the Barkin Index of Maternal Functioning
Time Frame: 3 months
Population: No data collected
Arm/Group | No Intervention: Usual Care Group | Experimental: Chabot Care Group
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Change in Maternal Confidence
Description: Measured by Maternal Confidence Questionnaire
Time Frame: 3 months
Population: No data collected
Arm/Group | No Intervention: Usual Care Group | Experimental: Chabot Care Group
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: Medication Adherence
Description: Measured by 1-item medication adherence questionnaire
Time Frame: 3 months
Population: No data collected
Arm/Group | No Intervention: Usual Care Group | Experimental: Chabot Care Group
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: 3 months]
Arm/Group | No Intervention: Usual Care Group | Experimental: Chabot Care Group
All-Cause Mortality (participants affected / at risk) | 0/15 | 0/16
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/16
Other Adverse Events (participants affected / at risk) | 0/15 | 0/16

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-05-19): https://cdn.clinicaltrials.gov/large-docs/89/NCT03990389/Prot_SAP_000.pdf